CLINICAL TRIAL: NCT05654779
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of CLL1-/CD33 Targeted LCAR-AMDR Cells Product in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CLL-1/CD33 Targeted LCAR-AMDR Cells in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Both the sponsors and collaborator are considering terminating the study
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022043
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-AMDR Cells Product (Experimental): Each subject will be treated with LCAR-AMDR Cells
  Interventions: Biological: LCAR-AMDR Cells Product

INTERVENTIONS:
Biological: LCAR-AMDR Cells Product — Subjects will receive a conditioning regimen before treatment with LCAR-AMDR cells

SUMMARY:
This is a prospective, single-arm, open-label, single dose-finding and dose-expansion study that evaluates the safety, tolerability, PK, and anti-tumor efficacy of LCAR-AMDR cells in subjects with relapsed/refractory Acute Myeloid Leukemia who received adequate standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in the clinical study; Fully understand and be Informed of the study and sign the Informed consent (Informed Consent Form, ICF)（For minors, the guardian shall also provide written informed consent ）; Willing to follow and able to complete all test procedures; Informed consent must be obtained before initiating any tests or procedures related to the study that are not part of the standard treatment of the subject's disease;
2. Age 14-60 years;
3. ECOG score: ≤2;
4. Relapsed/refractory AML must meet one of the following conditions:

   1. Twice or more relapse;
   2. Newly diagnosed AML patients who failed after 2 cycles of standard chemotherapy;
   3. Relapse within 12 months after CR, or relapse after 12 months with CR but failed to respond to conventional chemotherapy;
   4. Persistent extramedullary leukemia.
5. Meet the requirements of allogeneic HSCT
6. Expected survival ≥ 3 months;

Exclusion Criteria:

1. Subject with APL/AML-M3:t(15;17)(q22;q12)
2. Received any of the following treatments:

   * Previous allo-HSCT(Subjects who received allo-HSCT for more than 6 months, have stopped immunosuppressive drugs and have no active GvHD are not included in the exclusion criteria)
   * Previous gene therapy
   * Previous anti CD33/CLL1 therapy
   * Previous any target CAR-T cells therapy
3. Prior antitumor therapy with insufficient washout period;
4. CNS infiltration; Except for patients with prior CNS infiltration who are currently in remission;
5. HBsAg, HBV DNA, HCV-Ab, HCV RNA or HIV-Ab positive;
6. Pregnant or breast-feeding women;

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Time Frame: Minimum 2 years after LCAR-AMDR infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment
Recommended Phase 2 dose (RP2D) finding | 30 days after LCAR-AMDR infusion (Day 1)
  RP2D established through ATD+BOIN design
CAR positive T cells and CAR transgene levels in peripheral blood and bone marrow | 2 years after LCAR-AMDR infusion (Day 1)
  CAR positive T cells and CAR transgene levels in peripheral blood and bone marrow after LCAR-AMDR infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years after LCAR-AMDR infusion (Day 1)
  Objective Response Rate (ORR) is defined as the proportion of subjects who achieve CR or CRi after treatment via LCAR-AMDR cell infusion
Time to Response (TTR) | 2 years after LCAR-AMDR infusion (Day 1)
  Time to Response (TTR) is defined as the time from the date of first infusion of LCAR-AMDR to the date of the first response evaluation of the subject who has met all criteria for CR or CRi.
Duration of Response (DoR) | Minimum 2 years after LCAR-AMDR infusion (Day 1)
  Duration of Remission (DoR) is defined as the time from the first documentation of remission (CR or CRi) to the first documented relapse evidence of the responders
Event-free survival (EFS) | Minimum 2 years after LCAR-AMDR infusion (Day 1)
  Event-free survival (EFS) is defined as the time from the date of first infusion of the LCAR-AMDR to the first documented treatment failure, disease relapse or death (due to any cause), whichever occurs first
Overall Survival (OS) | Minimum 2 years after LCAR-AMDR infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LCAR-AMDR to death of the subject
The proportion of subjects who achieve CR or Cri and obtain bone marrow MRD negative. | Minimum 2 years after LCAR-AMDR infusion (Day 1)
  The proportion of subjects who achieve CR or Cri and obtain bone marrow MRD negative.
Incidence of anti-LCAR-AMDR antibody and positive sample titer | Minimum 2 years after LCAR-AMDR infusion (Day 1)
  Venous blood samples will be collected to measure LCAR-AMDR positive cell concentrations and the transgenic level of LCAR-AMDR, at the time points when anti-LCAR-AMDR antibody serum samples are evaluated

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad BoRen Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No